CLINICAL TRIAL: NCT06766942
Title: Effects of the Structured Sherborne Developmental Movement Program on Sensory and Motor Performance and Functional Status in Children With Autism Spectrum Disorders
Brief Title: Effects of the Sherborne Developmental Movement Program on Motor Performance in Children With Autism Spectrum Disorders
Acronym: absent
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Elif Dilan ATILGAN (Other)
Collaborators: Cukurova University (Other)
Responsible Party: Sponsor-Investigator, Elif Dilan ATILGAN, lecturer, Cukurova University
Organization: Cukurova University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2022/127; TDK-2023-16234 (Other Grant/Funding Number: Cukurova University Scientific Research Projects Unit)
Record Dates: First submitted 2025-01-04; First posted 2025-01-09 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Autism Spectrum Disorder
Keywords: autism spectrum disorder; motor activity; movement
MeSH Terms: conditions — Autism Spectrum Disorder; Motor Activity | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: An experimental study with 3 groups and a control group in which the effects of two independent variables were examined.
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- group in which the structured Sherborne developmental movement and sensory integration program was i (Experimental): The structured Sherborne developmental movement program and sensory integration program are implemented together.
  Interventions: Other: structured sherborne developmental movement program with sensory integration program
- the group to which the sensory integration program was applied (Experimental): only sensory integration program is applied.
  Interventions: Other: sensory integration program group
- control group (Other): Structured Sherborne developmental movement and sensory integration programs are not implemented.
  Interventions: Other: control group

INTERVENTIONS:
Other: structured sherborne developmental movement program with sensory integration program — In addition to the sensory integration therapy they receive at the rehabilitation center for 45 minutes, two days a week for 12 weeks, the Structured Sherborne Developmental Movement Program will be applied.
  Arms: group in which the structured Sherborne developmental movement and sensory integration program was i
Other: sensory integration program group — Sensory integration therapy programmed according to the individual's needs and disabilities will be applied to this group by an occupational therapist at the rehabilitation center for 45 minutes, 2 days a week for 12 weeks.
  Arms: the group to which the sensory integration program was applied
Other: control group — This group will not participate in any activities outside of the standard special education program.
  Arms: control group

SUMMARY:
The aim of this study was to investigate the effects of the Structured Sherborne Developmental Movement Program on sensory and motor performance and functional status in children with autism spectrum disorders.

DETAILED DESCRIPTION:
Autism is a complex disability that affects individuals differently, ranging from high-functioning to low-functioning autism. Autism is defined by cognition and observed behavior rather than specific medical diagnosis. It is a neurodevelopmental disorder classified in the category of pervasive disorders, characterized by impairment in socialization, unusual behaviors, and deficits in communication skills. In the United Kingdom alone, there are more than half a million people diagnosed with ASD, equivalent to 1 in every 100 people, and these numbers are rapidly increasing.

People with Autism Spectrum Disorder (ASD) tend to have similar characteristics and impairments in social skills, stereotypical behaviors (such as arm flapping), and unusual communication and interests. People with ASD tend to have poor social communication skills and lack a broad understanding of social cues. The effects of ASD put children at risk of remaining inactive, which can have harmful effects on their health.

In a study conducted by Pana et al., results show that students with ASD are not as physically active as their peers, but physical activity has a positive connection in promoting social interaction. A 2009 Estyn report showed that students demonstrated good development in their core skills through physical education, including problem-solving, working together, and listening, skills that could later be applied not only in physical education but also socially.

'Adapted physical education is the term used to describe services provided to school-age individuals from birth to 21 years of age.' Research has emphasized that when adapting lessons, children actively learn by teaching each other; it is important that all children, with and without disabilities, get this fundamental opportunity to coach each other.

The need for inclusive practice in physical education is now a crucial element in the national curriculum for students with special education, due to the recognition of psychological, physiological, and social benefits that physical education provides to students. The emphasis on inclusion in physical education has been largely recognized in recent years, especially for children with special educational needs.

Life skills learned in physical education can have significant effects on the learning of students with special needs, such as decreasing stereotypical behaviors and increasing adaptive behaviors. Children with autism struggle with movement skills, and their physical development may be delayed. Due to these physical and developmental deficiencies, teachers need to make adaptations in their lessons to ensure full participation of all students.

There are various barriers that autistic children face in physical education: anxiety, limited motor functionality, and overstimulation. If proper strategies and interventions are implemented, positive participation can be achieved, and children with autism can be encouraged to participate. Lang et al., in a study based on exercise activities for children with autism, found a decrease in stereotypical behavior and aggression, and an increase in adaptive behaviors such as focusing on lessons after physical activity.

The Sherborne Developmental Movement Method is an intervention created to develop motor movement for children with autism and severe learning difficulties. The main aim of the method is to develop general movement skills that enable children to overcome daily tasks rather than focusing on a sport. The Sherborne Developmental Movement Method can promote body awareness and relationships with others.

Veronica Sherborne's method is one of the most used methods in Europe and Poland in terms of developmental therapy. The fascinating aspect of this method is that those who use it approach the child in many ways while respecting the child's individuality. Both parents and children who actively participate in the lessons accept this method as a form of therapy.

Its adjustment to the needs and abilities of disabled children has enabled this method to be used as a therapeutic tool. In accordance with the method's principles, special emphasis is placed on the individual's psycho-physical development, communication, creativity, and changing behavior by participating in games. Games are the primary form of shaping contact with a child in terms of method.

The instructor, understood here as a guide, plays a very important role by a supporting person whose task in the developing movement method is to do exercises together with the person receiving therapy. This person should be the closest person who can guarantee a sense of security and stabilization, which is most often the mother. The basic principle of therapy is for the child to gain awareness of their own body parallel to their movement development.

When working with children with autism, its impact on emotional, social, and cognitive areas, the ease of adaptation of the method, and not requiring a large technical infrastructure have also contributed to the method's popularity among therapists. Another advantage is the participation of parents (presumably the child's parents) that allows some elements of the method to be used in a family.

There are various studies in the literature evaluating the effects of the Veronica Sherborne method on child development. Marchewka and Kowalska used the Bogdanowicz Behavior Observation Scale to conduct a preliminary analysis of the effectiveness of treatment according to the Veronica Sherborne method and evaluated changes in cognitive, emotional, social, and motor development of children with moderate intellectual disability, who had some autism features and attended kindergarten, compared to their healthy peers. It was found that lessons conducted according to the Sherborne Developmental Movement Method had the most beneficial effect on the development of emotional and cognitive areas and showed that the method was beneficial in the treatment of children with intellectual disabilities.

Błeszyński researched the effects of the Sherborne Method in children with ASD and found that this method was effective in autistic individuals and revealed the best effects when it came to the development of social and cognitive functions. He found that the method was particularly useful in working with young autistic children and children with autistic features (atypical autism in terms of time and level of intense autistic disorder). He also noted that the possibility of modifying and adapting the method according to the current needs and developmental abilities of participants was an additional advantage of the method, and for these reasons, it should be especially recommended to individuals working with children with ASD.

ELIGIBILITY:
Inclusion criteria:

Being between the ages of 6-12 Being diagnosed with autism spectrum disorder (ASD) Having the Family Consent Form approved by the child's primary caregiver Having the necessary prerequisite skills to participate in the study

* Being able to follow the commands given,
* Being able to imitate the model by taking the cues as a model,
* Having no other physical or mental disability other than ASD,
* Having no other health problems,
* Having the ability to hold the toilet.

Exclusion criteria:

Participant participating in an education and therapy program without the researcher's knowledge during the study Having problems adapting to the evaluation and education program Participant wanting to leave the study for any reason during the research process

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2025-01-09 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Bruininks-Oseretsky Test of Motor Proficiency-2 (BOT-2) | 3 months
  It was developed by Robert H. Bruininks and Brett D. Bruininks in 2005. It is a performance-based test that can be applied individually using engaging and targeted activities to evaluate a wide range of motor skills in individuals between the ages of 4-21. BOT-2 can be used for 5 different purposes, including supporting motor disorder diagnoses, screening, making placement decisions, evaluating and developing motor training programs, and conducting scientific research. BOT-2 consists of 4 sections: Fine Hand Control, Hand Coordination, Body Coordination, Strength, and Agility. Each section consists of two subtests and contains a total of 53 items. The total score to be obtained from the short form of BOT-2 is at least 0 and at most 88. It can be interpreted that motor performance increases as the score obtained from the short form increases.
Dunn Sensory Profile | 3 months
  The Dunn Sensory Profile, developed by Winnie Dunn in 1999, is a self-reported questionnaire that can measure children's sensory processing abilities and reveal the effects of sensory processing on children's functional performance in their daily lives, and can determine children's sensory performance in detail. The questionnaire can be applied to children with different types and degrees of disability. The assessment is carried out by rating the items in the questionnaire according to their frequency by the mother, father or caregiver; that is, the persons who are primarily responsible for the child's care. The questionnaire consists of 3 main sections, which are also divided into groups, and a total of 125 items.

SECONDARY OUTCOMES:
Gilliam Autistic Rating Scale-2 (GARS-2) | 3 months
  The Turkish version of the scale developed by Gilliam and adapted to Turkish culture by Diken, Ardıç, and Diken was used. The scale is a standardized tool for diagnosing, determining, and estimating the degree of ASD in individuals between the ages of 3-22. The scale is a 4-point Likert-type rating scale filled out by the caregivers of the individual (such as parents, teachers, caregivers). The scale can be used for screening and diagnosing individuals with ASD, evaluating severe behavioral problems, evaluating behavioral development, determining goals for individualized education plans, and collecting data for scientific studies. The scale consists of 3 subtests with 14 items in each subscale and a total of 42 items. The Autistic Disorder Index (ADI) score is calculated. As the AADI score increases, it can be interpreted that the degree of ASD increases.
Autism Social Skills Profile | 3 months
  The scale, developed by Bellini and Hopf in 2007 to determine the deficiencies experienced by children with autism in social skills, was adapted to Turkish by Demir in 2009 and named Autism Social Skills Profile-Turkish Form. The scale consists of 41 items and these 41 items are grouped under 3 factors. These factors are determined as "social reciprocity, social participation/avoidance and harmful social behaviors". The scale can be used with its three-factor subscales or as a single-factor form.
  The form filled out by parents of children diagnosed with autism between the ages of 6-17 uses a four-point Likert-type grading system. A high score obtained as a result of the scale evaluation indicates that the autistic child has positive social behaviors and social competence in terms of social functioning, while a low score indicates the opposite. However, reverse scoring is applied to 12 items defined as "harmful social behaviors" from the scale sub-dimensions.
Repetitive behaviors scale - revised - turkish version (TEDÖ-R-TV) | 3 months
  It is a clinical rating scale developed experimentally by Bodfish and his colleagues to evaluate repetitive behaviors and the severity of these behaviors. TEDÖ-R consists of six subscales, namely stereotypical behaviors (6 items), self-harming behaviors (8 items), compulsive behaviors (8 items), ritualistic behaviors (6 items), sameness/monotony behaviors (11 items), and limited interests (4 items), and a total of 43 items. This scale is filled out by interviewing the parents or directly by the parents. The items in the scale are scored on a four-point scale (0: No behavior, 1: Mild level, 2: Moderate level, 3: Severe level). As the score obtained from the scale increases, it is accepted that the severity of repetitive behaviors seen in children also increases.
Children's Sleep Habits Questionnaire (CSHQ) | 3 months
  This survey, which was created in 2000 for children regarding sleep patterns and problems, contains 33 questions. The survey includes eight subheadings: bedtime, difficulty falling asleep, amount of sleep, sleep anxiety, night waking, sleep problems, sleep breathing problems, and daytime sleepiness. There are 3 items for examining sleep routines (bedtime, time spent asleep throughout the day, time spent awake when awake at night). It is stated that the caregiver who can best observe the child should answer by considering the child's sleep habits from the previous week. The total score of all items is seen as 41 lines, and as this score increases, clinical significance emerges.
Quality of Life Scale for Children | 3 months
  It is a quality of life scale developed in 1999 to measure the health-related quality of life of children and adolescents aged 2-18. It consists of 4 subforms. These are physical health, emotional functioning, social functioning, and school functioning. Scoring is done in 3 areas. First, the total scale score, second, the total physical health score, and third, the psychosocial health total score, which is calculated by calculating the item scores that evaluate emotional, social, and school functioning. The items are scored between 0 and 100. If the answer to the question is marked as never, it gets 100 points, if it is marked as rarely, it gets 75 points, if it is marked as sometimes, it gets 50 points, if it is marked as often, it gets 25 points, and if it is marked as almost always, it gets 0 points. The higher the total scale score, the better the health-related quality of life is perceived.
Demographic Information Form | 3 months
  A short information form prepared by the researcher will be used to access demographic information about individuals with ASD.
Gastrointestinal Severity Index (GSI) | 3 months
  It is a scale used to determine the symptoms of the gastrointestinal system accompanying individuals with autism, with higher values paralleling the severity of symptoms. It includes questions about gastrointestinal symptoms such as constipation, diarrhea, stool consistency and odor, bloating and abdominal pain, unexplained daytime irritability and nighttime waking. Questions are scored as 0-1-2 and the total scale score is calculated as 15. Those with 3 and below are grouped as having low severity; those with more than 3 are grouped as having high severity gastrointestinal symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: ELİF D ATILGAN, Principal Investigator — Cukurova University
Locations (1):
- Cukurova University, Adana, Sariçam, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No